CLINICAL TRIAL: NCT05902377
Title: 68Ga-NY104 PET/CT Imaging in Patients With Confirmed or Suspicious Renal Cell Carcinoma
Brief Title: 68Ga-NY104 PET/CT Imaging in Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NYCR
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Renal Cell Carcinoma
Keywords: 68Ga-NY104; carbonic anhydrase IX
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NY104 PET/CT (Experimental): Each patient will receive one dose of 68Ga-NY104 by intravenous route. Dedicated whole-body PET/CT imaging will be performed.
  Interventions: Diagnostic Test: 68Ga-NY104 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-NY104 PET/CT — Participants will be administered a single, intravenous bolus of 68Ga-NY104 The recommended administered activity of 68Ga-NY104 is 1.8-2.2 MBq per kilogram bodyweight, subject to variation that may be required owing to variable elution efficiencies obtained during the lifetime of the 68Ga / 68Ga generator.
  The CT and PET imaging session will begin approximately 45 to 75 minutes after 68Ga-NY104 administration.
  Other Names: 68Ga-NYM005 PET/CT

SUMMARY:
This is a prospective, single-center study in patients with renal cell carcinoma. The goal is to determine the sensitivity and specificity of 68Ga-NY104 PET/CT in the detection of clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
Two types of patients will be recruited in this study. Type 1, patients with renal masses scheduled for surgery, type 2, patients with confirmed or suspicious recurrent/metastatic ccRCC. Each patient will receive one dose of 68Ga-NY104 by intravenous route. Dedicated whole-body PET/CT imaging will be performed. Imaging interpretations and reference standards will be used to estimate the sensitivity and specificity of 68G-NY104 PET/CT.

46 patients will be recruited in Peking Union Medical College Hospital. This study will be conducted according to local regulations and laws, the ethical principles that have their origin in the Declaration of Helsinki, and the principles of Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided for participation in the trial
2. Age ≥ 18 y
3. at least one of the following indications should be applied

   1. Scheduled for surgical resection of renal mass
   2. confirmed recurrent/metastatic clear cell renal cell carcinoma
   3. suspicion for recurrent/metastatic clear cell renal cell carcinoma

Exclusion Criteria:

1. On VEGF TKI treatment less than 1 week before 68Ga-NY104 PET/CT.
2. Pregnancy or lactation
3. Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Binary reading of focal lesions identified on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  Define lesion as PET positive or PET negative lesion.

SECONDARY OUTCOMES:
SUVmax of focal lesions identified on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  the tracer uptake is quantified using maximal standard uptake value (SUVmax) by drawing a 3-dimensional region of interest (ROI) over the lesion using a threshold of 40% SUVmax.

CONTACTS AND LOCATIONS:
Overall Officials: Huo Li, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu W, Zheng G, Yan X, Liu M, Li X, Cheng Y, Bai C, Zhang Y, Huo L. Diagnostic efficacy of [68Ga]Ga-NY104 PET/CT to identify clear cell renal cell carcinoma. Eur J Nucl Med Mol Imaging. 2024 Nov;51(13):4127-4133. doi: 10.1007/s00259-024-06801-y. Epub 2024 Jun 25. PMID 38916753